CLINICAL TRIAL: NCT07318597
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy, Safety, Pharmacokinetics, and Pharmacodynamic Effects of REGN13335, an Anti-PDGF-B Monoclonal Antibody, in Adults With Pulmonary Arterial Hypertension
Brief Title: Phase 2 Study of REGN13335 in Adult Participants With Pulmonary Arterial Hypertension (PAH)
Acronym: ILLUMINATE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R13335-PAH-2365; 2024-514754-79-00 (EU CTIS Number)
Record Dates: First submitted 2026-01-02; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Pulmonary Arterial Hypertension (PAH)
Keywords: Pulmonary Arterial Hypertension (PAH); Pulmonary Hypertension (PH); Elevated Pulmonary Vascular Resistance (PVR); World Health Organization (WHO) functional class II or III; Platelet-Derived Growth Factor-B (PDGF-B); REGN13335
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary

STUDY DESIGN:
Intervention Model Description: The study will include: A Double-Blind Treatment Period (DBTP) and an Open-Label Extension (OLE) period for participants who choose to continue treatment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- DBTP-Arm1 (Experimental)
  Interventions: Drug: REGN13335
- DBTP-Arm2 (Experimental)
  Interventions: Drug: REGN13335
- DBTP-Arm3 (Placebo Comparator)
  Interventions: Drug: Placebo
- OLE-Arm1 (Experimental)
  Interventions: Drug: REGN13335
- OLE-Arm2 (Experimental)
  Interventions: Drug: REGN13335

INTERVENTIONS:
Drug: REGN13335 — Administered per the protocol
  Arms: DBTP-Arm1; DBTP-Arm2; OLE-Arm1; OLE-Arm2
Drug: Placebo — Administered per the protocol
  Arms: DBTP-Arm3

SUMMARY:
This study is researching an experimental drug called REGN13335. The study is focused on participants with Pulmonary Arterial Hypertension (PAH). The aim of the study is to see how safe and effective REGN13335 is in participants with PAH who are taking other PAH medicines.

The study is looking at several other research questions, including:

* What side effects may happen from taking REGN13335
* How much REGN13335 is in the blood at different times
* Whether the body makes antibodies against REGN13335 (which could make REGN13335 less effective or could lead to side effects)

ELIGIBILITY:
Key Inclusion Criteria:

1. Documented clinical diagnosis of PAH (Group 1 PH according to the 7th World Symposium on Pulmonary Hypertension (WSPH))
2. WHO functional class II or III (slight to marked limitation of functional status due to PAH)
3. Receiving background Standard Of Care (SOC) therapy for PAH on a stable dose and regimen, as determined by the investigator, as described in the protocol
4. PVR ≥400 dynes∙sec/cm^5 (5 Wood units) based on Right Heart Catheterization (RHC) during the screening period
5. Has 6MWD ≥150 and ≤550 meters repeated twice during screening as described in the protocol

Key Exclusion Criteria:

1. Has Group 2 (PH associated with left heart disease), Group 3 (PH associated with lung diseases and/or hypoxia), Group 4 (PH associated with pulmonary artery obstructions), or Group 5 (PH with unclear and/or multifactorial mechanisms) PH according to the 7th WSPH
2. Pulmonary Arterial Wedge Pressure (PAWP) >15 mm Hg by RHC during the screening period
3. History of left-sided heart disease and/or clinically significant cardiac disease, as described in the protocol
4. Obstructive lung disease defined as Forced Expiratory Volume in 1 second (FEV1)/Forced Vital Capacity <0.7 and FEV1 <70% of the predicted value as described in the protocol
5. Evidence of interstitial lung disease as defined in the protocol
6. Evidence of chronic thromboembolic pulmonary disease or acute pulmonary embolism as described in the protocol
7. Participants requiring anticoagulation and/or antiplatelet therapy for an underlying medical condition as described in the protocol
8. Has any history of intracranial bleeding or any history of elevated intracranial pressure
9. Has any history of bleeding meeting criteria as described in the protocol

Note: Other protocol-defined Inclusion/ Exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2026-01-29 (Estimated); Primary Completion 2028-01-11 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Pulmonary Vascular Resistance (PVR) | At week 24

SECONDARY OUTCOMES:
Occurrence of Treatment-Emergent Adverse Events (TEAEs) | Through end of study, up to approximately 2.5 years
Severity of TEAEs | Through end of study, up to approximately 2.5 years
Change from baseline in circulating N-Terminal pro-B-type Natriuretic Peptide (NT-proBNP) concentrations | At week 24
Change from baseline in mean pulmonary artery pressure | At week 24
Change from baseline in cardiac output | At week 24
Change from baseline in cardiac index | At week 24
Change from baseline in right atrial pressure | At week 24
Change from baseline in 6-Minute Walk Distance (6MWD) | At week 24
Concentrations of functional REGN13335 in plasma | Through end of study, up to approximately 2.5 years
Concentrations of total soluble Platelet-Derived Growth Factor-B (PDGF-B) ligands in plasma | Through end of study, up to approximately 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/